CLINICAL TRIAL: NCT06486818
Title: Clinical Predictors of Short Term Outcomes of Ablation of Idiopathic Monomorphic PVCs
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Usama Mohammed Tony, Resident, Assiut University
Other Study IDs: Successful Pvcs ablation
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Arrythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ablation of idiopathic monomorphic PVCs — 3D carto ablation of idiopathic monomorphic PVCs

SUMMARY:
Clinical predictors of successful Pvcs ablation

DETAILED DESCRIPTION:
Clinical predictors of short term outcomes of ablation of idiopathic monomorphic pre mature ventricular contractions

ELIGIBILITY:
Inclusion Criteria:

* patients with idiopathic monomorphic PVCs

Exclusion Criteria:

* patients with heart failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 18 - 70
Sampling Method: Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical predictors of short term outcomes of ablation of idiopathic monomorphic PVCs | 2 years
  Successful Pvcs ablation

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes